CLINICAL TRIAL: NCT05538871
Title: Body Structure and Capacity Evaluation of Adults With Scoliosis
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00089305
Record Dates: First submitted 2019-05-03; First posted 2022-09-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Scoliosis
Keywords: Scoliosis; Degenerative scoliosis; Idiopathic scoliosis; Adult scoliosis; ICF; Deficits
MeSH Terms: conditions — Scoliosis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Degenerative scoliosis: Diagnosis of degenerative (De novo) scoliosis,
  Interventions: Diagnostic Test: Survey + Physical exam
- Adult idiopathic scoliosis: Diagnosis of idiopathic scoliosis,
  Interventions: Diagnostic Test: Survey + Physical exam
- Degenerative scoliosis - matched controls: Population sample matched to the degenerative scoliosis group.
  Interventions: Diagnostic Test: Survey + Physical exam
- Idiopathic scoliosis - matched controls: Population sample matched to the idiopathic scoliosis group.
  Interventions: Diagnostic Test: Survey + Physical exam

INTERVENTIONS:
Diagnostic Test: Survey + Physical exam — Survey:
  Demographic data Pain Oswestry disability index International Physical Activity Questionnaire Scoliosis Research Society (SRS-22r) Spinal appearance questionnaire Fear Avoidance and Beliefs Questionnaire Short Orebro musculoskeletal pain questionnaire Work Ability Index
  Physical exam:
  Repeated movements (MDT) Posture ROM Neuro Updated treatment based classification tests Pathoanatomical classification tests

SUMMARY:
Adults with scoliosis have not been the focus of much research in physical therapy despite their prevalence being very important. Adults with idiopathic scoliosis have a reported prevalence of about 2-11%. This includes adolescents with idiopathic scoliosis who have become adults but still have a scoliosis. They do not get much treatment as the adolescent treatment focuses on preventing worsening of the curvatures and the risk of progression is significantly reduced once a person reaches skeletal maturity. Still some patients experience self-image, function and pain issues which may be amenable to treatment using specific exercises as was recently shown. With ageing population a growing number of adults with de novo degenerative scoliosis is observed. This is a spinal misalignment due to spine degeneration. Adult degenerative scoliosis with pain is thought to affect about 24% of the ageing adults. This population has not been investigated very much.

Before planning conservative treatments for adults with scoliosis it would be important to describe what deficit these adults present that may be targeted by physical therapy. The objective of this study is to compare samples of patients with adults degenerative scoliosis, adult idiopathic scoliosis to matched healthy controls (for age, height and weight). Participants will complete questionnaires and a physical exam to identify which limitations they present that may be amenable to treatment with physical therapy. This information will assist planning trials to address the needs of these two neglected patient populations.

DETAILED DESCRIPTION:
Study design: A cross sectional study will be undertaken.

Participants will complete 45 minutes of questionnaires online using REDCAP then complete a physical exam for 1h15 including assessment of the posture, flexibility of the spine and lower extremity, neurological function, response to pain provocation test of the spine, pelvis and hips and tests of pulmonary function.

Sample size: A 0.8 point difference is expected between the expected score in the healthy groups (of 4.5) and the score in the scoliosis groups (expected scores of 3.7) on the SRS 22 with an expected SD of 1 in each group. With alpha=0.0167 (corrected for multiple comparisons) and beta=0.8 using an unilateral test needed 27 patients per group for a paired t test analysis.

Assessment methodology: Participants will bring their last X-ray and will fill out a survey and have a physical exam.

-Analysis : The population will be described with averages and standard deviations for the continuous data and frequencies with confidence intervals for the categorical.

Comparisons between groups: the continuous data among the 3 groups will be compared with paired and unpaired t test using Bonferroni post hoc comparison. Categorical data will be compared between groups with a Chi2 test (2 by 2).

References (see uploaded protocol).

ELIGIBILITY:
Inclusion criteria for the idiopathic scoliosis group :

* Diagnosis of idiopathic scoliosis
* Age ⩾18 years old
* Curve severity over 10°
* Fluent in English.

Inclusion criteria for the degenerative scoliosis group :

* Diagnosis of degenerative (De novo) scoliosis
* Age ⩾45 years old
* Curve severity over 10°
* Fluent in English.

Exclusion criteria for the scoliosis groups :

* History of spine surgery or
* History of diseases affecting the torso or lower extremity function
* Surgery or trauma
* Secondary scoliosis
* Unable to fill out the questionnaires or attend the physical examination,
* Pregnant or gave birth between 0 and 2 years ago.

Inclusion criteria for healthy groups:

* Age ⩾ 18 years
* Matched for age/height/weight (+/-5 years; +/- 10 lbs; +/- 10cm) to a scoliosis participant
* Fluent in English

Exclusion criteria for healthy groups:

* Serious systemic pathology
* Spine deformity
* Spine surgery
* Pregnant or gave birth between 0 and 2 years ago
* Unable to fill out the questionnaires or attend the physical examination
* Received treatments for the spine/the lower limbs within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults with adult idiopathic or degenerative scoliosis consulting a surgeon.
  All adults from the healthy/untreated population
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Socliosis Research Society 22-revised total score | baseline
  The SRS-22r is a quality of life questionnaire which consists of 22 questions assessing 5 quality of life domains: Function, Pain, Self-Image, Mental health (5 questions), satisfaction (2 questions). Each category is rated on 5. The categories are summed and divided by 5 to have a total score on 5 points. 5 is the best score and 1 the worst

SECONDARY OUTCOMES:
Pain intensity: Numerical rating scale | baseline
  Numerical rating scale from 0 to 10 where 0 is no pain and 10 the Worst imaginable pain. The patient has to select between: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. The value will be recorded separately for thoracic pain, lumbar pain and leg pain at the best, worse and current levels over the last 24 hours. All these scores are averaged for a total score.
Response to the Mechanical Diagnosis and Therapy (McKenzie) exam | baseline
  A repeated movement exam according to MDT will be completed to note centralisation, peripheralization , and detect directional preference. The patient will be asked to perform 10 repeated movements in flexion, extension, lateral side glides direction and the participant will be asked to report if symptoms became more proximal (centralisation), more distal (peripheralization) better or worse or if there was no change after the repetitions. The direction identified as providing centralization or the best pain response will be identified as the directional preference.
Perceived appearance | baseline
  The Spinal Appearance Questionnnaire (SAQ) consists of 11 pictogram questions and 12 multiple choice questions and an open question to assess the perceived appearance. A perceived appearance score (10-50) and an expectation score 4-20 will be calculated by averaging relevant items. A low score indicate good perceived appearance /50 and expectation /20.
Fear avoidance related to work and physical activity | baseline
  Fear Avoidance and Beliefs Questionnaire (FABQ). The FABQ was developed on the basis of the assumption that fear-avoidance beliefs play a major role in LBP-related disability. It comprises 16 items scored by the patient and includes sub-scores for fear-avoidance beliefs regarding work (0-42) and physical activity (0-24). A higher score indicates more strongly held fear avoidance beliefs.
Function | baseline
  Oswestry Disability Index (ODI). The ODI uses 10 questions with 5 answer options to assess the degree of disability associated with spinal disorders. The total score is out of 100 starting with 0. High score indicate high disability.
LBP prognosis score | baseline
  The modified Orebro Musculoskeletal Pain questionnaire (short version) is a 12 items questionnaire which assess pain and psycho social factors. 100 is the worst score and 0 the best.
Perceived ability to work | baseline
  Work Ability Index is a 5 items questionnaire which assess the perceived ability to work. 38 is the best and 5 the worst.
Physical activity level | baseline
  The International Physical Activity Questionnaire (short) assesses the time spent per the participant to do different level of physical activity during a week in minutes. The time spent at each activity levels is converted to a MET score for the each patient. High MET indicate more physical activity was performed.
Posture | baseline
  Photographies with landmarks: Posture photographs of the front and back and side profile of the participants will be collected to later extract the Posterior and Anterior Trunk Symmetry Indices (POTSI and ATSI). A plumbline and a flexicurve are used to assess the curves. High POTSI and ATSI scores indicate large deformity. High kyphosis and lordosis indices indicate hyperkyphosis and lordosis respectively.
Range of motion (lumbar, thoracic, lower limbs) | baseline
  Inclinometer to measure Range of motion in degree, the measurement of the lumbar flexion, extension and lateral flexion between T12L1 and S1 and the measurement of the thoracic flexion, extension and lateral flexion will be captured in degrees with double inclinometer technique between C7T1 and T12L1. The hip flexion is measured with the inclinometer on the front part of the tight. The straight leg raise and the prone knee bend test are measured with the single inclinometer on the front part of the ankle in both techniques. Higher degree readings indicate higher range of motion for all movements recorded with inclinometer (s).
Range of motion (Hip abduction, thoracic rotation) | baseline
  Goniometer in degree. The range of each hip abduction is recorded by the goniometer. Higher degree readings indicate higher flexibility. The range of thoracic rotation between a 2 meters stick and the lateral edge of the table is recorded to the nearest degree with a goniometer to indicate full spine rotation. Higher ranges indicate more flexibility.
Range of motion (lumbar rotation) | baseline
  Back Range Of Motion tool will be used to measured the degree or lumbar rotation available in the lumbar spine. Higher degrees indicate more flexiblity.
Sensory capacity | baseline
  Pic/Touch sensation on the lower limbs for each dermatome from L1 to S1. The examiner assesses for each dermatome if the participant discriminate most of the time the pic and the touch sensation or not. The front hip, front tight, medial knee, medial ankle, dorsal part of the big toe, heel, and the back of the knee are tested. Responses are recorded for each dermatomes on each side as can discriminates most of the time, does not discriminate most of the time and does not fell contact.
Voluntary motor capacity | baseline
  Strength of the lower limbs for each myotome from L1 to S1 measures with a dynamometer in pounds. The higher the score is higher the strength is. The hip flexion, knee extension, foot flexion/extension/eversion, and big toe extension are tested.
Involuntary motor capacity | baseline
  Patellar and Achilles Reflexes (hypereactive/hyporeactive/normal) are tested with an reflexe hammer. Reported as hyper, hypo or normal.
Nerves tension tests | baseline
  Prone Knee Bend (PKB) (knee flexion in a prone position) and Straight Leg Raise (SLR) (hip flexion with the knee extended in a supine position) tests. We recorde the range of motion in degree with the inclinometer and whether pain is produced pain or not by these tests.
Spirometric respiratory capacity | baseline
  Spirometer volumes (in liters): vital capacity, forced expiratory vital capacity, forced expiratory vital capacity after 1 sec (FEV1), FEV1 in % of maximal vital capacity. Flows (Liter/Sec): Maximal expiratory flow, Maximal expiratory flow at 25, 50, 75 % of the vital capacity, maximal inspiration flow. Higher are the volumes and flow better it is.
Flexibility | baseline
  The Beighton score is a 9 point score which assess general flexibility of the limbs (the examiner searches for any hyperextension of the elbows and the knees, the ability to touch the floor with the palms (knee extended), maximal 5th finger extension exceeding 90 dgegrees and ability to touch the forarm with the thumb. 9 is hypermobile, 0 is normal.
Prevalence of patients per potential treatment | baseline
  Prevalence in each of the treatment based classification algorithm classification: manipulation, stabilisation, specific exercise. The classification is based on the clinical findings described in the other outcomes and the algorithm is followed to classify if possible the participants in these 3 treatment categories (cf Fritz Subgrouping Patients With Low Back Pain: Evolution of a Classification Approach to Physical Therapy 2007 JOSPT)
Prevalence of patient in each specific LBP categories | baseline
  Patho-anatomical classification: Disc, disc+nerve root involvement, sacro iliac joint, spinal stenosis, spondylolisthesis. The research team classify (if possible) the participant in one of the categories based on the exam clinical findings(other outcomes listed above). Clinical criteria presented in Clinical classification in low back pain: best-evidence diagnostic rules based on systematic reviews by Petersen et al in 2017 are used to inform classification decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Parent, PT, PhD, Pr, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Faculty of Rehabilitation Medicine, Dept. Physical Therapy, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT05538871/Prot_SAP_000.pdf